CLINICAL TRIAL: NCT07276984
Title: Photobiomodulation Effect on Vietnamese Orthodontic Patients: A Randomized Clinical Trial
Brief Title: Photobiomodulation Effect on Vietnamese Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thanh Thuy-Nhat Cao, Principal, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22230-DHYD
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Root Resorption; Orthodontic; Tooth Movement
Keywords: photobiomodulation; pain; toothmovement; cumulative effect; LED; rootresoption
MeSH Terms: conditions — Agnosia; Root Resorption; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham LED device (Placebo Comparator): Patients wore the sham LED device without charging case for 10 minutes daily (5 minutes for the maxillary arch and 5 minutes for the mandibular arch at the same time each day). Patients did not know that LED device could emit light.
  Interventions: Device: Placebo LED device
- 850nm LED device (Experimental): Patients wore the LED device which emit near-infrared ligth at 850nm wavelength for 10 minutes daily (5 minutes for the maxillary arch and 5 minutes for the mandibular arch at the same time each day. Patients did not know that LED device could emit light.
  Interventions: Device: LED device

INTERVENTIONS:
Device: LED device — LED device emits near-infrared ligth at 850nm wavelength.
  Arms: 850nm LED device
Device: Placebo LED device — Sham LED device contains no charging case (emiting no light)
  Arms: Sham LED device

SUMMARY:
Since most orthodontic cases endure for 2 to 3 years or longer, patients are at a high risk of inflammatory root resorption and prolonged orthodontic pain, which is a common and unwanted side effect of their treatment. Photobiomodulation therapy utilizing light-emitting diodes (LEDs) offers a non-pharmacological approach for pain management, acceleration of tooth movement, and reduction of root resorption risk.

This randomized, placebo-controlled clinical trial aims to evaluate the effects of LED photobiomodulation on pain alleviation, acceleration of tooth movement, and mitigation of root resorption risk during orthodontic treatment. A total of 16 Vietnamese participants, aged 11 to 30 years, receiving fixed orthodontic treatment were randomly assigned to either an intervention group (LED therapy) or a control group (placebo). Patients were assessed at four consecutive follow-up visits at monthly intervals. Canine movement was measured by superimposing patients' 3D scans collected at the four follow-ups in 3D Slicer. At each visit, their pain intensity was measured using the Visual Analog Scale (VAS) to establish the baseline for that follow-up (0 hour), and then measured again at 24 hours and 48 hours post-visit. Furthermore, during each visit, the investigator collected patients' saliva and gingival crevicular fluid (GCF) to extract dentin sialoprotein (DSP), a biomarker of root resorption in humans.

The primary outcome is the difference in pain assessments between the intervention and control groups, the mobility of canines across groups, and the concentration of dentin sialoprotein in gingival crevicular fluid and saliva.

DETAILED DESCRIPTION:
During the orthodontic treatment period, patients must endure various discomforts, such as the risk of inflammatory root resorption and frequent pain, which typically occur due to the body's inflammatory response to the applied forces. Pain is commonly managed with non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen; however, these medications may induce adverse effects and potentially inhibit tooth movement. Photobiomodulation (PBM) therapy using light-emitting diodes (LEDs) has emerged as a non-pharmacological approach that may reduce pain, enhance tooth movement, and lower the risk of root resorption.

The objective of this randomized, placebo-controlled clinical trial is to evaluate the effects of LED PBM on pain reduction, enhancement of tooth movement, and mitigation of root resorption risk during orthodontic treatment. Sixteen participants aged 11 to 30 years undergoing fixed orthodontic treatment were randomly assigned to either the intervention group or the placebo group. In the intervention group, patients used the LED device for 10 minutes per day (5 minutes for the upper arch and 5 minutes for the lower arch) every day. In the placebo group, patients used a sham LED device (without a charging case) following the same procedure, 10 minutes per day. Patients in both groups were blinded to the light status while wearing the device. After finishing the aligning and leveling stage with Nickel and Titanium (NiTi) arch wires, during the phase of canine distalization with stainless steel arch wires, patients were assessed at four consecutive follow-up visits, scheduled at monthly intervals.

Canine movement was measured by superimposing sequential 3D digital scans obtained over these four visits using 3D Slicer software. Saliva and gingival crevicular fluid (GCF) samples were collected at each follow-up visit to measure dentin sialoprotein (DSP), a biomarker of root resorption in humans. Additionally, at each visit, patients' pain intensity was measured using the Visual Analog Scale (VAS) to establish the baseline for that follow-up (0 hour), and then measured again at 24 hours and 48 hours post-visit. The primary outcomes are differences between groups in canine displacement, pain intensity, and DSP concentration in both saliva and GCF.

The findings of this study may support the clinical application of LED PBM as a safe, non-invasive, and drug-free adjunctive therapy to improve patient comfort and reduce treatment-related risks during orthodontic care, particularly in Vietnamese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 11-30 years old who were required to undergo extraction of four premolars for orthodontic purposes.
* Four canines erupted in both arches.
* No active caries, no gingivitis, or periodontal disease was diagnosed through clinical examination and panoramic X-ray.
* No history of previous orthodontic treatment.
* No abnormality in tooth shape, number, or size.

Exclusion Criteria:

* Patients who smoked, had systemic diseases, and/or were using medications that could affect pain sensation.
* Patients who are diagnosed with severe root resorption based on their panorama X-ray image.

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Dentin sialoprotein (DSP) levels in saliva and gingival crevicular fluid | Pre-treatment, Baseline, 1-month follow-up, and 2-month follow-up.
  The primary endpoint is the difference in dentin sialoprotein (DSP) levels between the LED photobiomodulation group and the placebo group. DSP concentrations will be extracted from saliva and gingival crevicular fluid samples collected at four prespecified time points:
  * Pre-treatment
  * Baseline (initiation of canine distalization)
  * 1-month follow-up
  * 2-month follow-up DSP levels will be measured using Enzyme-Linked Immunosorbent Assay (ELISA). The primary comparison is the mean change in DSP levels across the follow-up period between the intervention and placebo groups, to evaluate the biomarker response associated with orthodontically induced inflammatory root resorption.
Rate of canine distalization (mm/month) compared across monthly intervals | Baseline to 1-month, 1-month to 2-month, and 2-month to 3-month intervals.
  Canine movement will be measured in millimeters by superimposing three-dimensional digital models of the maxilla and mandible. Digital models for participants in both study groups will be collected at the following visits:
  * Baseline (initiation of canine distalization)
  * 1-month follow-up
  * 2-month follow-up
  * 3-month follow-up
  Measurements will be performed using 3D Slicer software. The primary endpoint is the difference between the LED photobiomodulation group and the placebo group in the amount of canine movement observed during each monthly interval:
  * Baseline to 1-month
  * 1-month to 2-month
  * 2-month to 3-month
Change in pain intensity (VAS scores) | Immediately (0 hour) at Baseline, 1-month, 2-month, and 3-month follow-up visits.
  Pain intensity will be measured using a 100-mm Visual Analog Scale (VAS), illustrated as a 100mm ruler on questionnaire papers, where 0 represents no pain and 100 represents the worst imaginable pain. The primary endpoint is the difference in mean VAS scores between the LED photobiomodulation group and the placebo group. VAS scores will be recorded immediately at the time of each clinical visit. Measurements will be collected at four prespecified visits:
  * Baseline (initiation of canine distalization)
  * 1-month follow-up
  * 2-month follow-up
  * 3-month follow-up

SECONDARY OUTCOMES:
Time to peak pain intensity | 0 hour, 24 hours, and 48 hours after treatment initiation at Baseline, 1-month, 2-month, and 3-month visits.
  Time to peak pain intensity is defined as the time point (0 hour, 24 hours, or 48 hours) at which each participant records the highest Visual Analog Scale (VAS) score following initiation of canine distalization. Assessments will be performed at four scheduled visits: Baseline, 1-month, 2-month, and 3-month follow-up. The outcome will compare the proportion of participants whose peak pain occurs at each time point between the LED photobiomodulation group and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh TN Cao, MSc, Principal Investigator — University of Medicine and Pharmacy in Ho Chi Minh city
Locations (1):
- Faculty of Dentistry, University of Medicine and Pharmacy in Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The results of my primary outcomes including VAS scores of intervention and control groups
Supporting Information: Study Protocol
Time Frame: Start day: October 2025 End day: October 2027
Access Criteria: Students and researchers. Through my email address, thanh.caothuynhat@gmail.com